CLINICAL TRIAL: NCT02942823
Title: Kids Obesity Prevention Program Part 2 (KOP-2)
Brief Title: Kids Obesity Prevention Program Part 2
Acronym: KOP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Science Campus Tuebingen (Unknown); Department of School Psychology, University of Tuebingen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KOP_2
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2016-10

CONDITIONS: Obesity; Child
Keywords: obesity; child; primary prevention; serious game; nutrition; physical activity; psychosocial; stress; knowledge; diet; energy density; beverages; food pyramide
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Children in a primary school, aged between 9 and 12 years, play the serious game (two sessions, duration of each session 35 minutes, within two weeks). Additionally, the intervention group will take the game home on a tablet computer to play it with their parents in between session 1 and 2. The game equips the children and their parents with knowledge about the core areas nutrition, physical activity, and psychosocial factors.
  Interventions: Other: The serious game "KOP"
- Control (No Intervention): Children in a primary school, aged between 9 and 12 years, play the serious game (two sessions, duration of each session 35 minutes, within two weeks). The game equips the children with knowledge about the core areas nutrition, physical activity, and psychosocial factors. The parents are not involved.

INTERVENTIONS:
Other: The serious game "KOP" — The serious game transfers knowledge about nutrition (food pyramid, energy density of foods, which foods contribute to satiety and which not, energy in liquids, self-reflexive diagnostic tool to analyze daily food intake), physical activity (a motion-control to navigate through the game is partly used, relationship between energy expenditure and energy intake) and psychological aspects (relaxation-exercises, what is stress, stress-coping strategies).
  Arms: Intervention

SUMMARY:
Obesity and its associated comorbidities are becoming a key and rapidly growing public health problem. The cause of obesity is an imbalance between energy intake and energy expenditure in favor of the former. Childhood and adolescence are seen as critical time for its development. It is therefore crucial to provide both prevention and treatment actions already during childhood. The prevention and treatment weight-management programs in children focus on improving diet, eating behaviours, psychosocial aspects and increasing physical activity. One important basic requirement for any weight-management program is, that both children and their families are motivated and ready for change. Video games, including exergames, serious games or combined approaches offer additional chances in the treatment and prevention of obesity by approaching children in their environment and motivating them to deal with life-style topics.

As children do not decide alone what they eat - but their parents - the involvement of parents in the intervention appears to be very important to reach a sustained effect.

The investigators developed a motion-controlled serious game for children aged between 9 and 12 years, addressing all the three core areas nutrition, physical activity, and psychosocial factors. In addition to the motion control, a tablet is used for knowledge-based and cognitive tasks. In comparison to other studies the nutrition part not only deals with the food pyramid but also with the energy density of foods and liquids and offers a self-reflexive diagnostic tool to analyse daily food intake. Moreover, psychological aspects, especially stress and stress-coping strategies are addressed e.g. by relaxation-exercises and a reflexion exercise about leisure behaviour. The game consists of two sessions, having each a duration of about 35 minutes.

The aim of the KOP-1 study was to evaluate the game regarding its acceptance and efficacy in a cluster-randomized controlled trial in a primary school setting in children aged 9 to 12 years. The aim of the here presented KOP-2 study is to evaluate the game regarding its acceptance and efficacy in a randomized controlled trial in parents of primary school children aged 9 to 12 years receiving the KOP-1 intervention. Therefore, 4th grade pupils of the same school will be randomly allocated to an intervention and a control group. Both groups will play the game within two weeks, whereas the intervention group will take the game home on a tablet computer to play it with their parents in between session 1 and 2. At baseline, one day after session 2 and at four weeks follow-up, measurements will be performed in pupils and the parents of the intervention group. The primary outcomes of the study are the gain of knowledge (nutrition, psychosocial aspects) in parents and children, measured by a self-constructed questionnaires tailored specifically for the serious game. Secondary outcomes are the interaction of pupils and their parents for the intervention group, acceptance of the game, changes of nutrition behaviour, physical activity and intentions of the children to follow a healthy lifestyle, measured by mostly validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* all children which belong to the 4th graders of a primary school and their parents

Exclusion Criteria:

* children and their parents with massive linguistic difficulties will be excluded (after study participation; due to ethical reasons we can not do this ahead)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Knowledge of the parents about nutrition and psychosocial aspects by a self-developed questionnaire specific for the serious game | Change between baseline and intervention end, on average 4 weeks after baseline measurement
Knowledge of the children about nutrition and psychosocial aspects by a self-developed questionnaire specific for the serious game | Change between baseline and intervention end, on average 4 weeks after baseline measurement

SECONDARY OUTCOMES:
Interaction of pupils and their parents for the intervention group by a self-developed questionnaire tailored for this study | At the end of intervention, on average 4 weeks after baseline measurement (intervention group only)
Acceptance of the serious game by the parents using a self-developed questionnaire specific for the serious game | At the end of intervention, on average 4 weeks after baseline measurement (intervention group only)
Nutrition Score (Ernährungsmusterindex) by Kleiser et al., 2007 used in the KIGGS cohort (Studie zur Gesundheit von Kindern und Jugendlichen in Deutschland) | Change between baseline and four weeks follow-up
  Parents and children are independently asked to report the food frequencies for key foods in order to calculate the Ernährungsmuster index
Food frequency of specific foods which are addressed in the serious game | Change between baseline and four weeks follow-up
  Parents and children are independently asked to report the food frequencies of specific foods
Physical activity using a validated questionnaire filled in by the children and also the parents | Change between baseline and four weeks follow-up
  Parents and children are independently asked to fill in the questionnaire
Intentions of children to stick to a healthy lifestyle by using a tailored questionnaire specific for the contents of the serious game | Change between baseline and end of intervention, on average 4 weeks after baseline measurement

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Zipfel, Prof., Principal Investigator — University Hospital Tuebingen, Tuebingen, Germany